CLINICAL TRIAL: NCT02630017
Title: Motivated Behavior in Adults With and Without ADHD
Acronym: MOBE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 207259; Pro00068353 (Other: Duke University)
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: There are two parallel arms of this study (ADHD or non-ADHD subjects).
  Within each arm, each subject will be exposed to placebo and a drug (each at a different timepoint in the study). Although all subjects will receive both placebo and the drug, the order of presentation of the placebo and drug is counterbalanced across subjects (i.e., approximately half will receive the drug first and approximately half will receive the placebo first).
  For both study arms, regardless of whether the placebo is received first or second, the outcome measure will be calculated as the number of high effort selections.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADHD group (Experimental): Adults with ADHD
  Interventions: Drug: ADHD methylphenidate first, placebo second; Drug: ADHD placebo first, methylphenidate second
- non-ADHD group (Experimental): Adults without ADHD
  Interventions: Drug: Non-ADHD methylphenidate first, placebo second; Drug: Non-ADHD placebo first, methylphenidate second

INTERVENTIONS:
Drug: ADHD methylphenidate first, placebo second — double-blind, counter-balanced administration
  Arms: ADHD group
Drug: ADHD placebo first, methylphenidate second — double-blind, counter-balanced administration
  Arms: ADHD group
Drug: Non-ADHD methylphenidate first, placebo second — double-blind, counter-balanced administration
  Arms: non-ADHD group
Drug: Non-ADHD placebo first, methylphenidate second
  Arms: non-ADHD group

SUMMARY:
To investigate the effects of methylphenidate on motivated behavior in adults with and without ADHD

DETAILED DESCRIPTION:
This study has a mixed between- and within-subject design. Participants are young adults (aged 18-45) with ADHD and non-ADHD matched controls. They will be recruited from locations around the community, consented, screened for eligibility, then scheduled for 2 study days. Study days will be at least 48 hours apart. Thus, there will be a total of 3 lab visits across a 3 week period. Participants will be administered study drug on one study day and placebo on the other study day. They will complete a battery of cognitive/behavioral tasks and answer questionnaires on both study days.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy
2. between the ages of 18-45
3. non-ADHD subjects do not meet criteria for ADHD diagnosis or any subtype as determined by the Conners Diagnostic Interview or any T-Score > 55 on Inattentive Symptoms, Hyperactive-Impulsive Symptoms, Total Symptoms or ADHD Index subscales of the CAARS.
4. ADHD subjects meet criteria for a primary diagnosis of ADHD, any subtype, based on DSM-5

Exclusion Criteria:

1. inability to attend all required experimental sessions
2. significant health problems (e.g., current and uncontrolled liver, lung, or heart problems, current or past seizure disorder, serious head trauma)
3. primary diagnosis of Axis I psychiatric disorders other than ADHD (e.g., depression, anxiety disorder, schizophrenia)
4. meet DSM-5 criteria for substance use disorder other than nicotine in the past 12 months
5. use of psychoactive medications in the past 6 months as indicated by self-report
6. positive urine drug screen for drugs or positive breath alcohol concentration
7. contraindications for MPH
8. among women, nursing or a positive pregnancy test
9. IQ < 80 on Kaufman Brief Intelligence Test, 2nd edition
10. allergy to lactose
11. hypertension (If subject is ≤ 40 years of age and has blood pressure over 135/85 or heart rate over 90 beats per minute. If subject is > 40 years of age and has blood pressure over 130/80 or heart rate over 88 beats per minute)
12. body mass ratio > 30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, PhD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Addicott MA, Schechter JC, Sapyta JJ, Selig JP, Kollins SH, Weiss MD. Methylphenidate increases willingness to perform effort in adults with ADHD. Pharmacol Biochem Behav. 2019 Aug;183:14-21. doi: 10.1016/j.pbb.2019.06.008. Epub 2019 Jun 18. PMID 31226260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Within each study arm (ADHD or non-ADHD subjects), subjects were exposed to placebo and drug (each at a different timepoint in the study). Approximately half of the subjects within each arm received drug first and half received placebo first (i.e., order was counterbalanced).
Groups:
- ADHD Methylphenidate First, Placebo Second: Adults with ADHD who received drug (methylphenidate) first, followed by placebo
- ADHD Placebo First, Methylphenidate Second: Adults with ADHD who received placebo first, followed by drug (methylphenidate)
- Non-ADHD Methylphenidate First, Placebo Second: Adults without ADHD who received drug (methylphenidate) first, followed by placebo
- Non-ADHD Placebo First, Methylphenidate Second: Adults without ADHD who received placebo first, followed by drug (methylphenidate)
Period: Overall Study
Arm/Group | ADHD Methylphenidate First, Placebo Second | ADHD Placebo First, Methylphenidate Second | Non-ADHD Methylphenidate First, Placebo Second | Non-ADHD Placebo First, Methylphenidate Second
Started | 13 | 12 | 13 | 13
Completed | 12 | 11 | 11 | 12
Not Completed | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- ADHD: Adults with ADHD
- Non-ADHD: Adults without ADHD
- Total: Total of all reporting groups
Arm/Group | ADHD | Non-ADHD | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8) | 28 (7) | 31 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 18 | 12 | 30
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of High-effort Selections in the Effort-based Decision Making Task
Description: Number of high-effort selections in the effort-based decision making task from the placebo to the methylphenidate condition. This is a decision-making task where participants make high- or low-effort choices to earn a small financial reward. High-effort selections require 100 button presses with non-dominant hand pinky finger and low-effort selections require 30 button presses with dominant hand index finger (within 15 seconds). The number of high effort selections are summed across 50 trials of the task. This task measures the willingness to perform effort in relation to changing reward magnitude and probability. This is a basic science experiment, the clinical and/or physiological relevance of these results are not established.
Time Frame: 1 hour post drug (or placebo) administration for each study session
Population: Approximately half of the subjects within each arm (ADHD or non-ADHD) received drug first and half received placebo first (i.e., order was counterbalanced). The study was powered to compare two groups (ADHD vs non-ADHD). Since order of drug was counterbalanced, this means all ADHD subjects were evaluated under both placebo and drug conditions, and this is also true for the non-ADHD subjects.
Measure: Mean (Standard Error); unit: Number of high-effort selections
Groups:
- ADHD Subjects, Placebo Condition: Adults with ADHD, under the placebo condition
- ADHD Subjects, Methylphenidate Condition: Adults with ADHD, under the methylphenidate (drug) condition
- Non-ADHD Subjects, Placebo Condition: Adults without ADHD, under the placebo condition
- Non-ADHD Subjects, Methylphenidate Condition: Adults without ADHD, under the methylphenidate (drug) condition
Arm/Group | ADHD Subjects, Placebo Condition | ADHD Subjects, Methylphenidate Condition | Non-ADHD Subjects, Placebo Condition | Non-ADHD Subjects, Methylphenidate Condition
Number analyzed (Participants) | 23 | 23 | 23 | 23
Number of high-effort selections | 16.4 (2.2) | 21.35 (1.9) | 20.45 (2.2) | 19.8 (1.9)

ADVERSE EVENTS:
Time Frame: For each individual participant, 3 weeks (up to 60 days maximum)
Description: Data are being reporting according to the participant flow for the study.
Arm/Group | ADHD Methylphenidate First, Placebo Second | ADHD Placebo First, Methylphenidate Second | Non-ADHD Methylphenidate First, Placebo Second | Non-ADHD Placebo First, Methylphenidate Second
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT02630017/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT02630017/SAP_001.pdf